CLINICAL TRIAL: NCT00282334
Title: A Comparison of Telemedical and Conventional Antihypertensive Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Erling Bjerregaard Pedersen, Dept. of Medical Research, Holstebro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED.RES.2004.01.LBM
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Hypertension
Keywords: Telemedicine; Blood pressure; Quality of life; Cost-effectiveness
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home blood pressure telemonitoring (Experimental)
  Interventions: Device: Telemedical blood pressure monitoring
- Conventional blood pressure monitoring (No Intervention)

INTERVENTIONS:
Device: Telemedical blood pressure monitoring — Measurement of home blood pressure, three times per week for three months and once a week for three months.
  Arms: Home blood pressure telemonitoring

SUMMARY:
The aim of the study is to compare telemedical antihypertensive treatment based on home blood pressure monitoring and conventional antihypertensive treatment based on monitoring of blood pressure in the doctor's office.

We want to test the hypotheses that telemedical treatment is more effective in lowering blood pressure, provide better quality of life and is more cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* age 20 - 80 years
* office blood pressure > 150/95 mmHg or systolic blood pressure >150 mmHg and diastolic blood pressure < 90 mmHg

Exclusion Criteria:

* not able to perform home blood pressure measurements
* low compliance
* abuse of alcohol/ medicine
* unwillingness to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2004-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Line B Madsen, MD, Principal Investigator — Dept. of Medical Research, Holstebro Hospital, 7500 Holstebro, Denmark; Erling B Pedersen, Professor, Study Chair — Dept. of Medical Research, Holstebro Hospital, 7500 Holstebro, Denmark
Locations (1):
- Dept. of Medical Research, Holstebro Hospital, Holstebro, Denmark

REFERENCES:
- [Derived] Madsen LB, Christiansen T, Kirkegaard P, Pedersen EB. Economic evaluation of home blood pressure telemonitoring: a randomized controlled trial. Blood Press. 2011 Apr;20(2):117-25. doi: 10.3109/08037051.2010.532306. Epub 2010 Nov 24. PMID 21105759

RESULTS

PARTICIPANT FLOW:
Groups:
- Telemonitoring: Telemonitoring of home blood pressure
- Conventional: Conventional blood pressure monitoring
Period: Overall Study
Arm/Group | Telemonitoring | Conventional
Started | 113 | 123
Completed | 105 | 118
Not Completed | 8 | 5
Not completed — Withdrawal by Subject | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Blood Pressure Monitoring | Telemonitoring of Home Blood Press | Total
Number analyzed (Participants) | 123 | 113 | 236
Age Continuous [Mean (Standard Deviation); unit: years] | 55.0 (11.7) | 56.7 (11.6) | 55.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 58 | 117
  Male | 64 | 55 | 119
Region of Enrollment [Number; unit: participants]
  Denmark | 123 | 113 | 236

OUTCOME MEASURES:

1. Primary Outcome: Difference in Number of Patients Who Reached Target Blood Pressure
Time Frame: 6 months
Reporting Status: Not Posted
Measure: Number; unit: participants

2. Primary Outcome: Difference in Mean Daytime Systolic Ambulatory Blood Pressure From Baseline to Follow-up After Six Months
Description: Comparison of mean change in daytime systolic ambulatory blood pressure from baseline to follow up after 6 months between the two groups
Time Frame: baseline and 6 months
Population: Number of participants determined by power calculations. Analysis based on the principle of intention to treat with LOCF in cases missing at follow up.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Conventional Blood Pressure Monitoring | Telemonitoring of Home Blood Press
Number analyzed (Participants) | 123 | 113
mm Hg | -11.9 (14.8) [-6.1 to 1.5] | -9.6 (14.7) [-6.1 to 1.5]

ADVERSE EVENTS:
Arm/Group | Conventional Blood Pressure Monitoring | Telemonitoring of Home Blood Press
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/113
Other Adverse Events (participants affected / at risk) | 0/123 | 0/113

LIMITATIONS AND CAVEATS:
Technical difficulties with telemedical equipment,referral bias,unblinded study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes